CLINICAL TRIAL: NCT07362901
Title: A Prospective Study of Discomfort Symptoms in Patients With Aortic Disease After
Brief Title: Effects of Precise Education on Postoperative Discomfort Symptoms in Patients With Aortic Disease Undergoing Endovascular Intervention: a Single-center Randomized Controlled Study
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT20250170C-R1
Record Dates: First submitted 2025-12-12; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Aortic Dissection Aneurysm; Aortic Dissection Rupture; Aortic Dissection Involving the Descending Thoracic Aorta
Keywords: Nursing care; Postoperative complication management
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients with a Precise patient education involves distributing illustrated manuals that explain the specific circumstances related to six dimensions: surgical procedures, pain management, early mobilization, preoperative preparations, and potential discomfort symptoms.ortic dissection who received endovascular treatment
  Interventions: Behavioral: postoperative precise education
- 2: Routine nursing education involves distributing illustrated manuals to explain surgical procedures, pain management, early mobilization, preoperative preparations, and other relevant topics.

INTERVENTIONS:
Behavioral: postoperative precise education — Whether to implement precise education
  Groups: 1

SUMMARY:
The incidence and severity of post-procedural discomfort were evaluated in patients undergoing endovascular repair for aortic dissection across six symptom-related dimensions: immobilization-related issues, puncture site discomfort, adhesive-induced skin reactions, post-stent implantation syndrome, impairment in self-care ability, and physical/psychological stress responses.

DETAILED DESCRIPTION:
In this study, a customized postoperative discomfort symptom assessment questionnaire was developed based on patient-reported outcomes, with the objective of systematically evaluating common discomfort symptoms experienced by patients with aortic disease after endovascular intervention. The questionnaire covers six core dimensions: immobilization-related discomfort, puncture site-related discomfort, adhesive-related skin reactions, post-stent implantation syndrome, decline in self-care ability, and psychosomatic stress responses. Each symptom within these dimensions was scored on a 0-4 scale according to severity: 0 indicates no symptoms; 1 indicates mild symptoms that are tolerable; 2 indicates moderate symptoms that affect daily life but remain tolerable; 3 indicates severe symptoms requiring medical intervention; and 4 indicates extremely severe symptoms that are intolerable and require emergency treatment.

Pain was evaluated using the Numeric Rating Scale (NRS). Skin reactions such as lesions, blisters, bruises, erythema, and rashes were quantified by measuring the longest and widest dimensions of the lesion using a flexible measuring tape. Self-care ability was assessed using the Activities of Daily Living (ADL) scale combined with patient self-evaluation, focusing on four aspects: changing clothes, controlling bowel and bladder function, eating and drinking, and turning in bed.clothes, controlling bowel and bladder, eating and drinking, and turning in bed. Scoring ranged from 0 to 4, where 0 represented no impact, 1 represented mild impact, 2 indicated moderate impact (partial assistance needed but most activities completed independently), 3 indicated severe impact (major assistance needed, only a few activities independently completed), and 4 indicated almost complete loss of self-care ability.

Sleep disturbances were also rated from 0 to 4: 0 for no impact; 1 for mild disturbance with ability to fall asleep without special treatment; 2 for moderate disturbance, requiring a quiet environment to fall asleep; 3 for severe disturbance needing sleep medications; and 4 for complete inability to sleep. Abnormal sweating was similarly rated from 0 to 4: 0 for no sweating; 1 for slight perspiration; 2 for sweating in multiple areas such as armpits and back; 3 for soaked clothes or bed linens once; and 4 for soaking more than once.

Each discomfort dimension was clinically defined with clear inclusion criteria. Immobilization-related discomfort referred to symptoms resulting from postoperative limb immobilization, such as lower back soreness, which typically resolved after the immobilization was lifted. Puncture site-related discomfort was caused by pressure bandaging or sandbag compression, and included local pain, itching, bruising, erythema, or rash around the puncture site (excluding complications such as hematoma or pseudoaneurysm). Adhesive-related skin reactions included blisters, erosions, rashes, redness, itching, and bruising due to the use of pressure bandages or adhesive dressings.

Aortic disease-related discomfort symptoms included postoperative chest tightness, new chest or back pain different from the initial presentation, and abdominal bloating or pain (after excluding cardiovascular or gastrointestinal causes), which may be related to post-stent inflammatory responses or systemic stress. Decline in self-care ability referred to reduced independence compared to the preoperative state, including inability to change clothes independently, difficulty with toileting in bed, impaired eating or drinking, and inability to turn over in bed. Psychosomatic stress responses involved changes in psychological and physical states not present before surgery, such as sleep disturbances, fear of movement due to anxiety about puncture site bleeding, and profuse sweating.

Through this questionnaire, we aim to quantify patients' subjective discomfort from multiple dimensions in a systematic manner, providing a foundation for optimizing perioperative nursing interventions, improving patient comfort, and promoting enhanced recovery after endovascular treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with thoracoabdominal aortic disease
2. Patients who underwent endovascular treatment of the thoracoabdominal aorta via the femoral artery approach

Exclusion Criteria:

1. Aortic disease caused by infection
2. Aortic disease caused by trauma
3. Aortic disease treated by open abdominal surgery
4. Presence of systemic diseases uncontrollable by current medical standards (e.g., severe cardiac, pulmonary or hepatic dysfunction; advanced malignancy; cachexia; refractory severe coronary artery disease symptoms; coagulation disorders caused by genetic diseases, etc.)
5. Patients who have undergone endovascular aortic treatment via femoral artery access prior to this procedure due to other diseases (not related to the current aortic disease)
6. Patients with intracerebral hemorrhage, symptomatic stroke, myocardial infarction, or gastrointestinal bleeding within the past 6 months; patients under 18 years old; or those who refuse to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with aortic dissection undergoing endovascular treatment
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Immobilization-Related Score | Perioperative
  The immobilization-related score is used to assess the degree of discomfort resulting from limb immobilization implemented for medical purposes. Major symptoms include lower back soreness, lower back pain, back soreness, and back pain. The score ranges from 1 to 10, with higher scores indicating more severe immobilization-related discomfort.
Puncture Site-Related Score | perioperative
  The puncture site-related score is used to evaluate the degree of discomfort at and around the puncture site following transfemoral endovascular intervention. Main manifestations include pain around the puncture site, local erythema, and puncture site-related pseudoaneurysm, hematoma, or bleeding. The score ranges from 1 to 10, with higher scores indicating more severe puncture site-related discomfort.
Medical Adhesive-Related Skin Injury (MARSI) Score | perioperative
  The MARSI score is used to assess the severity of adverse skin reactions caused by the use of medical adhesive products or devices (e.g., catheter fixation tapes, dressings, compression bandages). Manifestations include blistering, skin breakdown, pain, erythema, and pruritus. The score ranges from 1 to 10, with higher scores indicating more severe skin injury.
Aortic Disease-Related Score | perioperative
  The aortic disease-related score is used to evaluate the degree of discomfort following endovascular aortic repair attributable to surgical manipulation, implanted devices (e.g., stents or stent grafts), or the progression of aortic pathology itself. Main symptoms include chest tightness or discomfort, chest or back pain, abdominal distension, and abdominal pain. The score ranges from 1 to 10, with higher scores indicating more severe aortic disease-related discomfort.
Self-Care Ability-Related Score | perioperative
  Based on Orem's self-care theory, the self-care ability-related score is used to assess the extent of impaired self-care resulting from physiological, psychological, or social limitations. Major aspects include difficulty with dressing and personal hygiene, restricted toileting in bed, impaired eating or drinking, inability to turn over independently, and negative impact on personal social image. The score ranges from 1 to 10, with higher scores indicating more severe self-care ability impairment.
Psychosomatic Stress-Related Score | perioperative
  The psychosomatic stress-related score is used to assess the severity of psychosomatic stress responses induced by internal or external stressors such as disease, trauma, or psychological pressure. Manifestations mainly include sleep disturbances, fear of movement due to excessive concern about puncture site or wound bleeding, and excessive sweating beyond usual levels. The score ranges from 1 to 10, with higher scores indicating more severe psychosomatic stress.

SECONDARY OUTCOMES:
Length of hospital stay | perioperative
  Length of hospital stay from admission to discharge
Patient satisfaction score | perioperative
  Patient satisfaction score ranges from 1 to 10, with higher scores indicating greater patient satisfaction.
Observation of complications | perioperative
  Incidence of inguinal puncture site bleeding, hematoma, and pseudoaneurysm

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol